CLINICAL TRIAL: NCT02980315
Title: A New Efficient EBV AssociatedTechnologies of T Cells in Treating Malignant Tumors and Clinical Application
Brief Title: A New EBV Related Technologies of T Cells in Treating Malignant Tumors and Clinical Application
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-ky-o43
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: nasopharyngeal carcinoma; EBV related cancers
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — Immunotherapy, Adoptive

ARMS (2):
- CAR-T cells (Experimental): the group treat with CAR-T cells
  Interventions: Other: CAR-T cells
- placebo (No Intervention): the group treat with CAR-T cells

INTERVENTIONS:
Other: CAR-T cells — the patients treat with CAR-T cells
  Other Names: adoptive immunotherapy
  Arms: CAR-T cells

SUMMARY:
The purpose of this study is to evaluate the safety of the designed LMP1-CAR -T cells and determine whether the CAR-T cells are effective in the treatment of EBV associated malignant tumors.

DETAILED DESCRIPTION:
Half of the patients will treat with LMP1-CAR-T cells,while the other half will receive a placebo.During the time of the treatment ,we will supervise the side effect of treated group.At last we compare the survival rate and health condition of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nasopharyngeal carcinoma

Exclusion Criteria:

* •pregnant woman

  * severe autoimmune diseases
  * serious infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Locations (1):
- SecondNanjingMU, Nanjing, Jiangsu, China